CLINICAL TRIAL: NCT03499652
Title: A Multicenter Prospective Cohort Study on Neonatal Bacterial Meningitis
Brief Title: Neonatal Bacterial Meningitis Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Children's Medical Center (Other); Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: XH-17-017
Record Dates: First submitted 2018-04-08; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Bacterial Meningitis; Neonatal Infection
MeSH Terms: conditions — Meningitis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — cerebrospinal fluid, blood, urine, excrement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- derivation cohort: The data of derivation cohort are used to derive the neonatal bacterial meningitis risk score
  Interventions: Diagnostic Test: neonatal bacterial meningitis risk score
- validation cohort: The data of validation cohort are used to validate the neonatal bacterial meningitis risk score
  Interventions: Diagnostic Test: neonatal bacterial meningitis risk score

INTERVENTIONS:
Diagnostic Test: neonatal bacterial meningitis risk score — In the validation cohort,according to the neonatal bacterial meningitis risk score, we will suggest neonates who reach certain score to take a lumbar puncture, but we will not interfere with clinicians' decision

SUMMARY:
Neonatal bacterial meningitis (BM) is a devastating infection that occurs more commonly in neonates than in any other age group, and is associated with significant morbidity and mortality, especially in developing countries. In this study, we aimed to develop a clinical risk score model, according to the available clinical syndromes and commonly laboratory tests, for screening BM among full-term neonates in a large-scale retrospective cohort, and prospectively validated the risk score in multicenter cohort.

DETAILED DESCRIPTION:
In this study, we aimed to develop a clinical risk score model, according to the available clinical syndromes and commonly laboratory tests, for screening BM among full-term neonates in a large-scale retrospective cohort, and prospectively validated the risk score in multicenter cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a positive cerebrospinal fluid culture of bacterial pathogen(s)
* Subject has a positive blood culture of bacterial pathogen and counts of white blood cells in cerebrospinal fluid ≥ 20×106/L
* Subject has counts of white blood cells in cerebrospinal fluid ≥ 20×106/L and counts of neutrophils ≥ 10×106/L as well as suspected clinical symptoms

Exclusion Criteria:

* History of brain trauma, brain tumor, cerebral palsy, epilepsy, and ventricular shunt device
* History of accepting neurosurgery
* Subject has missing data

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Eligible participants were full-term neonates, aged older than 3 days, who were suspected with BM and received LPs.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
neonatal bacterial meningitis risk score | 1 day
  Our researchers grade the patients with the neonatal bacterial meningitis risk score to identify patients with bacterial meningitis, patients with risk score ≤ 3 points considered to be the low-risk group, and patients with risk score > 3.1 points considered the high-risk group, and the risk score model has no maximum or minimum value.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided
we plan to share all the individual participant data information available to our cooperative hospitals through emails